CLINICAL TRIAL: NCT05041140
Title: Hyperpolarized 129-Xenon Imaging in Adult Hematopoietic Cell Transplant Recipients With Pulmonary Impairment
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1170; NCI-2021-09252 (Other: NCI-CTRP Clinical Trials Processing Registry)
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary; Pneumonia; Hematopoietic System--Cancer
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: 29-XeMRI imaging — 129-XeMRI scan

SUMMARY:
This study is designed to measure the correlation of hyperpolarized 129-Xe magnetic resonance imaging (129-XeMRI) in allogeneic hematopoietic cell transplant (allo-HCT) recipients at MD Anderson Cancer Center (MDACC) who develop bronchiolitis obliterans syndrome (BOS) or BOS stage 0p (pulmonary impairment not meeting the definition for BOS, defined below) and controls with chronic graft-versus-host disease (cGVHD).

The primary objective of the study is to correlate 129-Xenon measures of ventilation, gas exchange, and pulmonary circulation with spirometric and quantitative CT measurements.

A secondary objective is to determine whether measurement of 129-Xe MRI characteristics in patients with BOS stage 0p can predict BOS progression 6 months after enrollment.

DETAILED DESCRIPTION:
The primary objective of the study is to correlate 129-Xenon measures of ventilation, gas exchange, and pulmonary circulation with spirometric and quantitative CT measurements.

A secondary objective is to assess the differences in 129-Xe MRI characteristics between patients with and without OS progression at 6 months after enrollment. Other secondary objectives include the assessment of the relationship of VDP, barrier defects (continuous variable), and circulation defects (continuous variable) with pulmonary function, quantitative CT measurements, SGRQ, and SF-6D.

ELIGIBILITY:
Inclusion Criteria:

- Allo-HCT recipients who are at least 18 years of age and have BOS (n=10 patients), BOS 0p (n = 10 patients), or cGVHD of a non-lung organ without evidence of pulmonary impairment (n = 5 patients).

Healthy Cohort - Inclusion Criteria:

We will perform only XeMRI imaging on 10 healthy adult (18 years and older) volunteers with no medical issues for technical calibration of the XeMRI technology. Members of the study team may serve as healthy volunteers if they have no prior history of lung disease. These data will not be included as part of the analysis.

Exclusion Criteria:

1. Participants unable to follow up at MD Anderson for routine clinical care
2. Inability or unwillingness to give informed consent
3. Relapsed disease or life expectancy less than 6 months at time of enrollment
4. Severe claustrophobia precluding MRI imaging
5. Active pulmonary infection
6. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Population
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
To correlate 129-Xenon measures of ventilation, gas exchange, and pulmonary circulation with spirometric and quantitative CT measurements. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ajay First Name: Ajay MI: Last Name: Degree: Organizational, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org